CLINICAL TRIAL: NCT06090409
Title: Assessing Dietary Patterns and Implementing Cost-effective Interventions to Encourage a Plant-based Diet in an Underserved Urban Population
Brief Title: Encouraging a Plant Based Diet in an Underserved Urban Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Oatly Group AB (Unknown)
Responsible Party: Principal Investigator, Erin Murphy, Assistant Professor, M.D., University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23.0126
Record Dates: First submitted 2023-03-17; First posted 2023-10-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Food Neophobia; Food Preferences; Dietary Habits
Keywords: Food Neophobia, Plant-based Diet
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Food Preferences; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free/Subsidized Community Supported Agriculture (CSA) produce along with education. (Experimental): Patients who self-elect to enroll in subsidized/free Community-supported agriculture produce shares will also receive Education on the benefits of a plant-based diet.
  Interventions: Other: Implementing free/subsidized agricultural produce to encourage a plant-based diet.
- Education Alone (Active Comparator): Patients will receive educational information about the benefits of plant-based eating.
  Interventions: Other: Implementing free/subsidized agricultural produce to encourage a plant-based diet.

INTERVENTIONS:
Other: Implementing free/subsidized agricultural produce to encourage a plant-based diet. — Providing educational material on the benefits of a plant-based diet, simple recipes, food swaps and free/subsidized produce.

SUMMARY:
The investigator's goal is to promote a plant-based diet amongst the underserved urban population of Louisville with the help of educational aids and the provision of affordable resources.

DETAILED DESCRIPTION:
Primary care clinic patients who screen positive for food insecurity between 2021-2023 will be eligible for this study (~200 patients). Patients will be recruited by one of four means: during standard clinic visits, or via phone, Electronic Medical Record message, or mail. Registry of patients will be de-identified and list of identifiers will be stored separately from the data set. Data will be stored on password protected computers only available to select research staff. Investigators will utilize a preamble in lieu of informed consent.

The primary outcome will be to measure the readiness of patients to adhere to a plant-based diet. Investigators will assess readiness using Food Neophobia inventory and will perform a brief Diet Inventory at simultaneous timepoints. Education surrounding benefits and easy ways to increase plant-based eating will be distributed to all participating patients. Enrollment in a local income-based subsidized Community Supported Agriculture share (weekly farm produce box during growing season) will be offered to all patients. Patients can opt into this service, and we will track which patients enroll. Before, during, and after the Community Sponsored Agriculture produce time period, Food Neophobia and Diet Inventory will be reassessed.

Adherence to plant-based eating between the patients who received access to subsidized food and education versus those who received education alone will be evaluated. Qualitative open-ended feedback will be obtained at all time points.

The secondary outcomes are to measure weight loss, reduction in blood pressure, and improvement in hemoglobin A1C and lipid profile wherever applicable.

Statistical significance is not attempting to be reached, but rather the associations between food neophobia and ability to change diet will be evaluated, as well as other qualitative open-ended feedback.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older screening as food insecure since 2021
* Patients willing to complete survey data

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Food Neophobia | 1 year
  Assess the readiness of participants to adhere to a plant-based diet while identifying potential barriers to the adhering to the diet.
Diet Inventory | 1 year
  Measure adherence to the plant-based diet between the education only group and the education + free/subsidized agricultural produce.

SECONDARY OUTCOMES:
Reduction in blood pressure | 1 year
  Systolic and diastolic blood pressure will be recorded when done per Standard of Care.
Improvement in lipid profile | 1 year
  measure of hemoglobin A1C will be recorded when done per Standard of Care.
Weight Loss | 1 year
  measure of weight will be recorded when done per Standard of Care.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Murphy, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Ambulatory Internal Medicine Resident Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient identifiers will be visible to Principal investigator and Co-Investigatory and kept in separate password-protected database. Other study investigators will see Individual Participant Data with identifiers removed.
Supporting Information: Study Protocol, SAP
Time Frame: entirety of study and for 1 year after